CLINICAL TRIAL: NCT03448913
Title: Prospective Observational Single-centre Study: Difference in the Incidence of Chronic Pain After Breast Surgery Between General Anesthesia and General Anesthesia Associated With PECS Block (Block REducing Pain After Surgery Trial)
Brief Title: Block REducing Pain After Surgery Trial
Acronym: BREAST
Status: Completed | Type: Observational
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Alessandro De Cassai, Medical Doctor, University of Padova
Other Study IDs: 4355/AO/17
Record Dates: First submitted 2018-02-19; First posted 2018-02-28 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Chronic Pain Post-Procedural
Keywords: Anesthesia, Regional ;PECS block

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PECS block+ General anesthesia: Patients undergoing mastectomy, partial mastectomy and/or axillary clearance who received PECS block AND general anesthesia for the surgery.
  Interventions: Procedure: PECS block
- General anesthesia: Patients undergoing mastectomy, partial mastectomy and/or axillary clearance who received general anesthesia only for the surgery.

INTERVENTIONS:
Procedure: PECS block — It consists in injection of 20-30 ml of local anesthetic between pectoral minor, pectoral major, and serratus muscles.
  Groups: PECS block+ General anesthesia

SUMMARY:
This observational study evaluates difference in chronic pain after six months from surgery between patients who received PECS block and general anesthesia versus general anesthesia alone.

DETAILED DESCRIPTION:
PECS block is used as a pain relief technique during breast surgery. However at the actual state of knowledge there is no strong evidence that its use could lower incidence of chronic pain compared to general anesthesia alone.

Moreover for its use an adequate skill with ultrasound machine is required. For this reason only some anesthesiologists in our reality use this technique it in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* programmed breast surgery
* informed consent

Exclusion Criteria:

* bilateral breast surgery

Ages: 18 Years to 86 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients needing breast surgery (mastectomy, partial mastectomy and/or axillary clearence)
Sampling Method: Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Chronic pain at six months | six months
  Presence of chronic pain at six months after surgery. For this purpose patient will be asked to report presence of pain on breast, neck, axilla or arm. If patient will report pain a further question about intensity (NRS) and quality (we will ask to patient to describe with words from one to three the pain). Furthermore we will ask to patient if he had take any action (eg drugs) to treat pain

SECONDARY OUTCOMES:
Chronic pain at three months | three months
  Presence of chronic pain at three months after surgery. For this purpose patient will be asked to report presence of pain on breast, neck, axilla or arm. If patient will report pain a further question about intensity (NRS) and quality (we will ask to patient to describe with words from one to three the pain). Furthermore we will ask to patient if he had take any action (eg drugs) to treat pain
Chronic pain at nine months | nine months
  Presence of chronic pain at nine months after surgery. For this purpose patient will be asked to report presence of pain on breast, neck, axilla or arm. If patient will report pain a further question about intensity (NRS) and quality (we will ask to patient to describe with words from one to three the pain). Furthermore we will ask to patient if he had take any action (eg drugs) to treat pain
Chronic pain at twelve months | twelve months
  Presence of chronic pain at twelve months after surgery. For this purpose patient will be asked to report presence of pain on breast, neck, axilla or arm. If patient will report pain a further question about intensity (NRS) and quality (we will ask to patient to describe with words from one to three the pain). Furthermore we will ask to patient if he had take any action (eg drugs) to treat pain
Difference in opioid consumption during surgery | day of surgery
  Difference in opioid consumption during surgery (Fentanyl as mcg/kg/h; Remifentanil as mcg/kg/min)
Difference in pain in the first 24 hours after surgery | first 24 hours after surgery
  maximum and mean NRS score in the first 24 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro De Cassai, MD, Principal Investigator — University of Padova
Locations (1):
- University of Padova, Padua, Italy

IPD SHARING:
Plan to Share IPD: Undecided
De.identified individual participant data for all primary and secondary measures will be probably be made available

REFERENCES:
- [Background] Cronin-Fenton DP, Norgaard M, Jacobsen J, Garne JP, Ewertz M, Lash TL, Sorensen HT. Comorbidity and survival of Danish breast cancer patients from 1995 to 2005. Br J Cancer. 2007 May 7;96(9):1462-8. doi: 10.1038/sj.bjc.6603717. Epub 2007 Apr 3. PMID 17406360
- [Background] Andersen KG, Kehlet H. Persistent pain after breast cancer treatment: a critical review of risk factors and strategies for prevention. J Pain. 2011 Jul;12(7):725-46. doi: 10.1016/j.jpain.2010.12.005. Epub 2011 Mar 24. PMID 21435953
- [Background] Macdonald L, Bruce J, Scott NW, Smith WC, Chambers WA. Long-term follow-up of breast cancer survivors with post-mastectomy pain syndrome. Br J Cancer. 2005 Jan 31;92(2):225-30. doi: 10.1038/sj.bjc.6602304. PMID 15655557
- [Background] Blanco R. The 'pecs block': a novel technique for providing analgesia after breast surgery. Anaesthesia. 2011 Sep;66(9):847-8. doi: 10.1111/j.1365-2044.2011.06838.x. No abstract available. PMID 21831090
- [Result] Wijayasinghe N, Andersen KG, Kehlet H. Analgesic and Sensory Effects of the Pecs Local Anesthetic Block in Patients with Persistent Pain after Breast Cancer Surgery: A Pilot Study. Pain Pract. 2017 Feb;17(2):185-191. doi: 10.1111/papr.12423. Epub 2016 Feb 9. PMID 26857336